CLINICAL TRIAL: NCT05710003
Title: Effect of Breathing Exercises and Upper Limb Endurance Exercises in Pregnant Women Presented With Physiological Dyspnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Entsar Hsanen (Other)
Responsible Party: Sponsor-Investigator, Entsar Hsanen, doctor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: breathing exercises pregnancy
Record Dates: First submitted 2023-01-25; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Pregnancy Related; Dyspnea
Keywords: dyspnea; breathing exercises; pregnancy
MeSH Terms: conditions — Dyspnea | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: This study will include pregnant ladies presented to respiratory outpatient clinic with physiological dyspnea at the third trimester of pregnancy
Masking Description: single group pf patients and follow up effect of breathing exercises and upper limb exercises in perceived dyspnea and quality of life(fatigue scores)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: breathing exercises — A-breathing exercises: 20 times per hour. While setting down, deep breathing is taken from the nose while mouth is closed, breath holding for at least ten seconds, then slow maximal exhalation for at least 10 seconds.
  B-Upper Limb Endurance Exercises (low weight and high repetition) : Study participants will be educated to perform upper limb exercises every 4 hours. Three exercises will be repeated 10×3 times with 1 minute rest in between.
  Breathing exercise and upper limb endurance exercises is explained in the reminder in details
  Other Names: upper limb endurance exercises

SUMMARY:
To evaluate the effects of breathing exercises and upper limb endurance exercises in pregnant women presented with physiological dyspnea

DETAILED DESCRIPTION:
Pregnant women undergo various anatomical and physiological changes so that they can cope with the increased physical and metabolic demands of their pregnancies. Cardiovascular, respiratory, haematological, renal, gastrointestinal and endocrine systems undergo important physiological adaptations needed to allow development of the fetus and to allow the mother and fetus to survive the demands of childbirth . On the other hand, dyspnea can be caused by pregnancy complications, thus requiring specific medical treatment. Shortness of breath is common during pregnancy, occurring in 60% to 70% of healthy pregnant women . The aim of the study is to evaluate the effects of breathing exercises and upper limb endurance exercises in pregnant women presented with physiological dyspnea

ELIGIBILITY:
1. Inclusion criteria: pregnant women presented with physiological dyspnea.
2. Exclusion criteria:

   1. Non physiological causes of dyspnea in pregnancy

      * Cardiac: arrhythmia, constrictive pericarditis , pericardial effusion , coronary heart disease , congestive heart failure , intracardiac shunt , cardiomyopathy , valvular heart disease.
      * Chest wall, pleura, lungs: bronchial asthma, bronchiectasis ,bronchiolitis ,chronic obstructive pulmonary disease, pulmonary emphysema, interstitial lung disease, sarcoidosis ,lung tumor narrowing or compressing the airways , pleural effusion , pulmonary right-to-left shunt , pulmonary hypertension ,elevated hemi diaphragm, phrenic nerve palsy, kyphoscoliosis
      * CNS and neuromuscular: amyotrophic lateral sclerosis , mitochondrial disease polymyositis/ dermatomyositis
      * Metabolic: renal failure , thyroid disease
      * Head and neck : laryngeal tumor ,vocal cord paralysis , vocal cord dysfunction , tumor compressing the upper airways , tracheal stenosis , goiter
      * Others: anemia , anxiety disorder, panic attacks, , ascites , obesity, abdominal wall hernia
   2. Refusal to participate

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Modified dyspnea Borg scale | 4 weeks
  Modified Borg Dyspnea Scale is most commonly used to assess symptoms of breathlessness. It has a range from 0 to 10 (with 0 being no exertion and 10 being maximum effort).

SECONDARY OUTCOMES:
Modified Medical Research Council Dyspnea Scale (mMRC) | 4 weeks
  allows the patients to indicate the extent to which their breathlessness affects their mobility.
  The 1-5 stage scale is used alongside the questionnaire to establish clinical grades of breathlessness.
London chest activity of Daily Living questionnaire (LCADL) | 4 weeks
  It consist of four domains Selfcare, domestic activities, physical activities and leisure activities.
  Selfcare, domestic, physical and leisure activities contains 4, 6, 2 and 3 items respectively. Each item is graded by numbers 0-5, 0 mean little or no dyspnea and 5 mean worst dyspnea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee SY, Chien DK, Huang CH, Shih SC, Lee WC, Chang WH. Dyspnea in pregnancy. Taiwan J Obstet Gynecol. 2017 Aug;56(4):432-436. doi: 10.1016/j.tjog.2017.04.035. PMID 28805596
- [Background] Hegewald MJ, Crapo RO. Respiratory physiology in pregnancy. Clin Chest Med. 2011 Mar;32(1):1-13. doi: 10.1016/j.ccm.2010.11.001. PMID 21277444
- [Background] Melzer K, Schutz Y, Boulvain M, Kayser B. Physical activity and pregnancy: cardiovascular adaptations, recommendations and pregnancy outcomes. Sports Med. 2010 Jun 1;40(6):493-507. doi: 10.2165/11532290-000000000-00000. PMID 20524714